CLINICAL TRIAL: NCT06479629
Title: The Effect of Piracetam on the Clinical Outcomes of Diabetic Patients with Peripheral Neuropathy
Brief Title: The Effect of Piracetam on Diabetic Peripheral Neuropathy Patients
Acronym: DPN
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: King Salman International university (Other)
Responsible Party: Principal Investigator, Hamsa Amr Mohamed Attia, Teaching Assistant at clinical pharmacy department, King Salman International university
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHCL 5611
Record Dates: First submitted 2024-06-16; First posted 2024-06-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetes; Peripheral Neuropathy; Piracetam
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases | interventions — Piracetam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Piracetam Group (Active Comparator): receiving standard care according to the institution's protocol, along with 800mg oral tablet of Piracetam three times every day for the whole duration of the study ( 3 Months) Standard care includes insulin therapy with or without oral hypoglycemics and vitamin b complex.
  Interventions: Drug: Piracetam
- Control Group (Placebo Comparator): will receive standard care in accordance with the institution protocol in addition to placebo for 3 months.
  Standard care includes insulin therapy with or without oral hypoglycemics and vitamin b complex.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Piracetam — 800mg oral tablet of Piracetam three times every day for 3 months
  Other Names: no other interventions
  Arms: Piracetam Group
Drug: Placebo — starch tablet
  Arms: Control Group

SUMMARY:
Aim of the work:

To evaluate efficacy and safety of Piracetam in Diabetic patients with peripheral neuropathy.

Scientific background:

Diabetes mellitus (DM) is known to precipitate various neurologic complications, with diabetic neuropathy (DN) emerging as a significant microvascular consequence affecting both type 1 and type 2 diabetes mellitus (T2DM) patients. Notably, diabetic neuropathy can manifest even at the onset of type 2 diabetes mellitus. Peripheral neuropathy stands as the most common subtype of diabetic neuropathy, impacting nearly half of all individuals with diabetes over their lifetimes, as per recent guidelines. The development of diabetic neuropathy (DN) involves various metabolic and cellular processes, including inflammation and oxidative stress. Inflammation, characterized by cytokines and inflammatory cells, plays a role in diabetic neuropathy progression. Reactive oxygen species (ROS) contribute significantly, with low levels of antioxidants exacerbating the condition. Accumulation of advanced glycation end products (AGEs) further damages nerves. diabetic neuropathy leads to significant pain and discomfort for patients, yet current treatments often fall short of expectations. Improving treatment strategies is crucial to relieve suffering and improve the well-being of those affected by diabetic neuropathy. Piracetam shows promise in managing diabetic neuropathy (DN) based on both preclinical and clinical studies. It may enhance central nervous system function by influencing neurotransmitter release, potentially alleviating diabetic neuropathy symptoms. Additionally, piracetam's neuroprotective properties could shield nerve cells from oxidative stress and inflammation, which are key contributors to diabetic neuropathy nerve damage.

DETAILED DESCRIPTION:
Ninety eligible patients will be randomly assigned to two groups:

A) Piracetam Group (45 patients) receiving standard care plus 800mg Piracetam tablets thrice daily for the study duration, and B) Control Group (45 patients) receiving standard care plus a placebo for 3 months. Standard care involves insulin therapy with or without oral hypoglycemics and vitamin B complex supplementation.

Baseline assessments will include age, weight, height, sex, race, baseline pain intensity, non-opioid analgesic use, diabetes medications, overall sleep quality, symptom duration, medication and medical histories, and laboratory tests such as HbA1c and fasting glucose levels. These assessments represent the outcomes of the clinical trial:

Pain intensity was measured using the McGill Pain Questionnaire. Vibratory sensation is assessed through the Michigan Neuropathy Screening Test (MNSI).

Quality of life was evaluated using the EQ-5D-5L questionnaire. Sleeping disturbances related to diabetic neuropathy were measured using the Pittsburgh Sleep Quality Index (PSQI).

Cognitive function was examined with the Montreal Cognitive Assessment Test (MoCA).

Serum biomarker levels of Brain-Derived Neurotrophic Factor (BDNF) measured. The safety and tolerability of piracetam were assessed throughout the study. These assessments will provide valuable insights into the efficacy and safety of piracetam in managing diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (>the age of 18).
2. Established diagnosis of type 2 Diabetes Mellitus.
3. Patients receiving insulin therapy.
4. Stable regimen for at least 3 months prior to inclusion in the study
5. HbA1C>7.5%

Exclusion Criteria:

* Patients with inadequate hepatic function Alanine aminotransferase, Aspartate aminotransferase (ALT, AST > or equal to 3 times upper normal limit).
* Patients with myopathy, epilepsy, malignancy, unstable psychiatric illness, bleeding tendency, or peripheral vascular diseases.
* Patients with an estimated Glomerular Filtration Rate (GFR) Less than 45 ml/min and albumin/creatinine ratio or urea to creatinine >30.
* Patients with any conditions that could confound pain assessment (for ex: other severe pain or skin conditions in the area affected by neuropathy.
* Cognitive or language difficulties that would impair understanding/completion of the assessment instruments.
* Presence of foot ulcers.
* Causes of neuropathy other than diabetes and significant neurological diseases.
* Pregnant and/or breastfeeding women.
* Use anticonvulsants, antidepressants, membrane stabilizers, and opioids.
* Patients with a history of Substance use and alcohol abuse,
* Patients with a history of (cerebral hemorrhage) or at risk of blood diseases.
* Patients allergic to piracetam

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of efficacy:1. Measurment of McGill Pain Scale: | 3 Months
  Neuropathic pain severity will be assessed at baseline and every 4 weeks during the whole study duration using The Short-Form McGill Pain Questionnaire (SF-MPQ).The SF-MPQ is a concise assessment tool consisting of 15 items that evaluate both the sensory and affective dimensions of pain experience, Participants rate the intensity of each item on a four-point scale ranging from 0 (none) to 3 (severe). By summing the intensity values for the corresponding descriptors, sensory (11 items), affective (4 items), and total (15 items) pain scores can be obtained.
Evaluation of efficacy: 2. Assessment of the vibratory sensation using Michigan neuropathy screening instrument | 3 Months
  Assessment of patients' vibratory sensation will be performed using Michigan Neuropathy screening Instrument , The MNSI consists of two parts, one of them a questionnaire for the patient, a higher score (with a maximum of 13 points) indicates a greater presence of neuropathic symptoms, and the second part is done by the examiner and contains physical examination tests, A high score on the questionnaire, reduced or absent vibration sense, reduced or absent ankle reflexes, and reduced or absent sensation on the monofilament test are all indicative of neuropathic symptoms, suggesting the presence of diabetic neuropathy. Patients who score above 2 points on a 10-point scale in the clinical section of the MNSI are considered to have neuropathic symptoms.
Evaluation of efficacy:3. Assessment of EQ-5D-5L Score: | 3 Months
  Assessment of patients' Quality of life will be performed using EQ-5D-5L questionnaire, The EQ-5D-5L consists of a concise descriptive system questionnaire and a visual analog scale (EQ VAS),The questionnaire captures a straightforward profile of an individual's health state, while the EQ VAS offers an alternative approach to gauge an individual's self-rated overall current health, The updated version of the EQ-5D, known as the EQ-5D-5L, introduces five levels of severity for each of the existing five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Within the EQ-5D-5L descriptive system, there are five dimensions, and each dimension encompasses five response levels, ranging from 1 which indicates absence of problems to 5 which indicates Inability to perform/extreme problems.
Evaluation of efficacy: 4. Assessment of Pittsburgh sleep quality index Score: | 3 Months
  Sleep disturbance will be assessed, The Pittsburgh sleep quality index questionnaire about usual sleeping habits for the past month only. These questions are consolidated to create seven distinct "component" scores, each with a scoring range of 0-3 points. It is important to note that a score of "0" indicates the absence of any difficulties, while a score of "3" signifies the presence of severe difficulties. Subsequently, the seven component scores are combined to generate a single "global" score, spanning from 0 to 21 points. Within this framework, a score of "0" indicates the absence of any difficulties across all domains, while a score of "21" signifies the presence of severe difficulties in all areas.
Evaluation of efficacy: 5. Measurment of Montreal Cognitive Assessment Scale | 3 Months
  Cognitive function will be assessed. The Montreal Cognitive Assessment (MoCA), which is a quick screening assessment used to detect elderly people who have mild cognitive impairment (MCI). It is a single-page examination that may be performed in 10 minutes. This test has a maximum score of 30, with a result of 26 or higher deemed normal. A score of less than 26 without associated functional impairment indicates a diagnosis of mild cognitive impairment. Furthermore, a score of less than 26 combined with functional impairment implies that dementia is in its early stages. It is worth mentioning that an additional point is given whether the individual has completed 12 years of formal education or less.
Evaluation of efficacy: 6. Evaluation of serum Brain-derived neurotrophic factor: | 3 Months
  Blood sample will be withdrawn from each patient at baseline and after 3 months and separated sera will be stored at -80 C till analysis. Serum Brain-derived neurotrophic factor will be assessed for each patient using ELISA kits.
7.Incidence of Adverse Events | 3 months
  Patients will be educated about any expected side effects and will be required to report any of them.

IPD SHARING:
Plan to Share IPD: No